CLINICAL TRIAL: NCT06239090
Title: Study of Brain Activations and Physiological Responses Using NeuroBiofeedback in Patients With Multiple Sclerosis.Study of Brain Activations and Physiological Responses Using NeuroBiofeedback in Patients With Multiple Sclerosis
Brief Title: Study of Brain Activations and Physiological Responses Using NeuroBiofeedback in Patients With Multiple Sclerosis
Acronym: NBF2023
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Giuseppa Maresca, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBF2023
Record Dates: First submitted 2024-01-09; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Multiple Sclerosis; Mood Disorders; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis; Mood Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (IG) (Experimental): During each session IG patients will view their recorded brain waves and physiological responses in a computer screen, while a professional will explain to them what they need to do to intervene and make corrective changes to their brain waves.
  Interventions: Device: Rehacor-T
- sham group (SG) (Sham Comparator): SG patients will be given irrelevant information (recorded data of other patients) and thus, they cannot modulate their cortical activation.
  Interventions: Behavioral: Sham Intervention

INTERVENTIONS:
Device: Rehacor-T — During each session of bio/neurofeedback IG patients will view their recorded brain waves and physiological responses in a computer screen, while a professional will explain to them what they need to do to intervene and make corrective changes to their brain waves.
  Arms: intervention group (IG)
Behavioral: Sham Intervention — SG patients will be given irrelevant information (recorded data of other patients) and thus, they cannot modulate their cortical activation and see only the scenarios
  Arms: sham group (SG)

SUMMARY:
Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system (CNS) characterized by inflammation, demyelination, gliosis, and neuronal loss. Neurological symptoms may include visual disturbances, numbness and tingling, focal weakness, bladder and bowel incontinence, and cognitive impairment. Some previous studies have indicated that the NeuroBiofeedback (NBF) technique could be a promising new treatment for the rehabilitation of many neurological disorders and neurodegenerative diseases, including MS. Several studies have investigated the beneficial effects of this technique on the motor and cognitive outcomes of MS, mainly aiming to evaluate motor performance, fatigue and chronic pain. Few studies have focused on the evaluation and treatment of cognitive processes with NBF, except for one study on information processing speed. Specifically, regarding the application of NBF techniques in MS, recent literature has demonstrated that modulation of the alpha-theta rhythm has led to an improvement in attentional processes with consequent reduction in anxiety. Therefore, the objective of this study is to verify the effectiveness of NBF training on the modulation of cortical activity and physiological responses through the exposure of subjects with MS to cognitive tasks and training for mood regulation.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system (CNS) characterized by inflammation, demyelination, gliosis, and neuronal loss. Neurological symptoms may include visual disturbances, numbness and tingling, focal weakness, bladder and bowel incontinence, and cognitive impairment. Some previous studies have indicated that the NeuroBiofeedback (NBF) technique could be a promising new treatment for the rehabilitation of many neurological disorders and neurodegenerative diseases, including MS. Several studies have investigated the beneficial effects of this technique on the motor and cognitive outcomes of MS, mainly aiming to evaluate motor performance, fatigue and chronic pain. Few studies have focused on the evaluation and treatment of cognitive processes with NBF, except for one study on information processing speed. Specifically, regarding the application of NBF techniques in MS, recent literature has demonstrated that modulation of the alpha-theta rhythm has led to an improvement in attentional processes with consequent reduction in anxiety. Therefore, the objective of this study is to verify the effectiveness of NBF training on the modulation of cortical activity and physiological responses through the exposure of subjects with MS to cognitive tasks and training for mood regulation.

Patients will not undergo an experimental procedure as foreseen by the study; the clinical and neuropsychological variables that will be collected for the study are those that are commonly collected by the neuropsychologist, in particular the main neuro-cognitive functions (memory, language, attention and executive functioning) and emotional abilities (meta cognition) will be considered. After enrollment, the clinical background and baseline characteristics of patients will be assessed. Enrolled patients will be randomly assigned to IG and SG. After randomization, patients will undergo instrumental examinations and neuropsychological evaluation, as required by the protocol. Patients in both groups will undergo 2 neurofeedback training sessions. All recruited subjects will be evaluated at two time-points: a first evaluation at baseline (T0) and at the end of the training (T1). Patients will undergo stimulation training via NBF 2 times a week for two months, for a total of 16 sessions. The procedure and execution of the training requires that the subjects are connected to a series of electrodes that will record the cortical electrical activity. During each session, IG patients will view their recorded brain waves and physiological responses in front of a computer screen, while a professional will explain to them what they need to do to intervene on what they see, in order to correctively modify their brain waves. While SG patients will be provided with irrelevant information (recorded data from other patients) and therefore will not be able to modulate their cortical activation

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years ;
* Confirmed clinical diagnosis;
* Written informed consent obtained from the patient;
* Moca score ≥ 20;
* Patients with no contraindications to perform MRI and EEG.
* Clinical stability
* documented absence of relapse in the last month before treatment

Exclusion Criteria:

* Ascertained diagnosis of multiple pathologies,
* Patients with severe psychotic symptoms;
* Epilepsy;
* Drug use;
* Endocrine-metabolic encephalopathies.
* Presence of multiple therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological assessment | 30 minutes
  For the neuropsychological evaluation, the Brief Repeatable Battery of Neuropsychological Tests is used, which measures cognitive deterioration in patients with multiple sclerosis. The test evaluates memory, attention and learning speed. The higher the score, the better the performance. Administration of the total test battery takes approximately 30 minutes.
Mood assessment | 15 minutes
  The Beck Depression Inventory is a self-report instrument, composed of 21 items that evaluate the cognitive symptoms, affective, motivational and somatic aspects of depression. Each item is rated on a Likert scale from 0 to 3 points. Scores between 0 and 13 indicate the absence of depressive symptoms; scores between 14 and 18 indicate mild-moderate depression; scores between 19 and 29 indicate moderate-severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy